CLINICAL TRIAL: NCT00495469
Title: A Once-Daily Dose-Ranging Study of GSK189075 Versus Placebo In The Treatment of Type 2 Diabetes Mellitus in Treatment-Naïve Subjects
Brief Title: Dose-Ranging Study In Subjects With Type 2 Diabetes Mellitus Who Are Treatment-Naive
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KG2110375
Record Dates: First submitted 2007-06-29; First posted 2007-07-03 (Estimated); Results first posted 2017-10-30 (Actual); Last update posted 2017-10-30 (Actual); Status verified 2017-09

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes mellitus HbA1c
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- GSK189075 (Experimental): Participants will receive GSK189075 for 12 weeks
  Interventions: Drug: GSK189075
- Placebo (Placebo Comparator): Participants will receive GSK189075 matching Placebo for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GSK189075 — GSK189075 is available as a white, capsule-shaped tablet dosage form containing 50mg, 125mg, 250mg or 500mg of GSK189075 per tablet
  Arms: GSK189075
Drug: Placebo — Available as Placebo matching tablet to GSK189075
  Arms: Placebo

SUMMARY:
This is a dose-ranging study to evaluate the efficacy, safety and tolerability of a range of doses of GSK189075 (an SGLT2 inhibitor) compared to placebo, administered over 12 weeks in treatment-naive subjects with type 2 diabetes mellitus

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a documented diagnosis of T2DM and HbA1c ≥7.0% and ≤9.5% measured by the central laboratory at Visit 1.

  * Note: Subjects with HbA1c <7.5% must have a fasting fingerstick glucose ≥7 mmol/L (126 mg/dL) at Week 0, prior to randomization.
  * Note: The proportion of subjects who are randomized with an HbA1c <7.5% will be limited to be no more than 20% (approximately 51 subjects)
* Subjects who are treatment-naïve, and have not taken insulin, or any oral or injectable anti-diabetic medication in the past 3 months and have not taken a glucose lowering agent for ≥4 weeks at any time in the past, or subjects who are newly diagnosed and treated with diet and exercise for a minimum of 6 weeks
* Subjects who are 18 to 70 years of age inclusive at the time of Screening.
* Females of childbearing and non-childbearing and potential are eligible to participate as follows:

  * Women of childbearing potential must be willing to use one of the following contraception methods: intrauterine device, condom or occlusive cap (diaphragm or cervical/vault caps) plus spermicidal agent for at least 30 days prior to the start of study medication, throughout the study and the follow-up visit. Note: use of oral contraceptives is not permitted.
  * Women of non-child bearing potential are defined as follows: females regardless of age, with functioning ovaries who have a current documented tubal ligation, or who are surgically sterile (i.e. documented total hysterectomy or bilateral oophorectomy), or females who are post-menopausal.

All females must have a negative urine pregnancy test on the day of, and prior to randomization.

* Informed Consent: a signed and dated written consent must be obtained from the subject before any procedures are performed.

Exclusion Criteria:

* Metabolic Disease

  * Diagnosis of Type 1 diabetes mellitus
  * History of ketoacidosis which has required hospitalization
  * Thyroid disorder
  * TSH <0.4 MIU/L (<0.4 MCIU/mL) or >5.5 mIU/L (>5.5 MCIU/mL) at Screening
  * BMI of <22 kg/m2 or >43 kg/m2
  * Significant weight gain or loss (as defined as >5% of total body weight) in the 3 months prior to Screening
* Diabetic Medication

  * Has taken insulin, or any oral or injectable anti-diabetic medication within 3 months of screening
  * Has taken insulin or any oral or injectable anti-diabetic medication ≥4 weeks at any time in the past
* Cardiovascular Disease

Recent history or presence of clinically significant acute cardiovascular disease including:

* Documented myocardial infarction in the 6 months prior to Screening.
* Coronary revascularization including percutaneous transluminal coronary angioplasty (PTCA) or coronary artery bypass graft (CABG) surgery either planned and/or occurred in the 6 months prior to Screening.
* Unstable angina in the 6 months prior to Screening.
* Clinically significant supraventricular arrhythmias requiring medical therapy, or history of nonsustained or sustained ventricular tachycardia. Symptomatic valvular heart disease or valvular heart disease requiring therapy other than endocarditis prophylaxis.
* Congestive heart failure (CHF, New York Heart Association (NYHA) Class II to IV) requiring pharmacologic treatment or the NYHA Class criteria in accordance with the local prescribing information for pioglitazone.
* Blood pressure (BP) >150/100mmHg. If a subject is receiving permitted antihypertensive therapy, then they must be on stable dose(s) of therapy for at least 4 weeks prior to Screening.
* Based on local readings, the subject has an initial QTc interval (Bazett's)≥450msec at Screening, and after two additional ECGs taken 5 minutes apart, the average of the QTC interval from the three ECGs is ≥450msec.
* Other clinically significant ECG abnormalities which, in the opinion of the Investigator, may affect the interpretation of efficacy or safety data, or which otherwise contraindicates participation in a clinical trial with a new chemical entity.
* Fasting triglycerides ≥400mg/dL (4.56mmol/L) at Screening. If a subject is receiving permitted lipid-lowering therapy, then they must be on a stable dose(s) of therapy for at least 6 weeks prior to Screening. Niacin and bile acid sequestrants are prohibited.

  * Hepatic Disease

Has a diagnosis of active hepatitis (hepatitis B surface antigen or hepatitis C antibody), or clinically significant hepatic enzyme elevation including:

Any one of the following enzymes greater than 2 times the upper limit of the reference range (ULRR) value at Screening.

* alanine aminotransferase (ALT)
* aspartate aminotransferase (AST)
* alkaline phosphatase (AP) Has a total bilirubin level that is >1.5 times the ULRR at Screening with the exception of suspected or confirmed Gilbert's disease.

  * Pancreatic Disease
* Secondary causes of diabetes:
* history of chronic or acute pancreatitis

  * Renal Disease

Significant renal disease at Screening as manifested by:

* Glomerular filtration rate (GFR) <60mL/min (as calculated by Quest at Visit using the Modification of Diet in Renal Disease (MDRD) equation

  •≥1+ protein on urine dipstick
* Trace or ≥1+ leukocyte esterase on urine dipstick
* Trace or ≥1+ blood on urine dipstick
* Positive nitrite on urine dipstick
* Recurrent genitourinary tract infections defined as ≥2 episodes of complicated or uncomplicated cystitis or pyelonephritis in the 6 months prior to Screening.

  * Concurrent Disease
* Has any concurrent condition or any clinically significant abnormality identified on the screening physical examination, laboratory tests (including blood electrolytes), ECG, including pulmonary, neurological or inflammatory diseases, which, in the opinion of the investigator, may affect the interpretation of efficacy and safety data, or which otherwise contraindicates participation in a clinical trial with a new chemical entity.
* History of significant co-morbid diseases active in the 6 months prior to Screening (e.g., cholecystitis, acute pancreatitis, gastrointestinal disease, chronic diarrhea, etc.).
* History of malignancy within the past 5 years other than superficial squamous cell carcinoma (non-invasive on pathology) or basal cell carcinoma (successfully treated with local excision).
* History of cervical cancer in situ treated definitively at least 6 months prior to Screening.

  * Concurrent Medication

Is currently taking or has taken any of the following medications in the 8 weeks prior to Screening:

* Digoxin
* Warfarin and other oral anticoagulants (aspirin and non-steroidal anti-inflammatory drugs are permitted)
* Bile acid sequestrants
* Niacin (excluding routine vitamin supplementation)
* Antiobesity agents (including fat absorption blocking agents)
* Oral or injectable corticosteroids (inhaled, topical and intranasal corticosteroids are permitted)
* Loop diuretics
* Monoamine oxidase inhibitors and tricyclic amines
* Antiretroviral drugs
* St John's Wort
* Oral chromium 9.Breast Feeding 10.Other
* Current smoker who is unable to abstain from smoking while in the clinic at each visit
* Has a history of alcohol or substance abuse within the past year at Screening or alcohol or substance abuse during treatment, as determined by the investigator:
* Unwilling to refrain from the use of illicit drugs and adhere to other protocol-stated restrictions while participating in the study
* Has an average weekly intake of alcohol of >21 units or an average daily intake of >3 units (males) or an average weekly intake of >14 units or an average daily intake of >2 units (females). One unit is equivalent to a half pint of beer or 1 measure of spirits or 1 glass of wine
* Has participated in any study with an investigational or marketed drug in the 3 months prior to Screening.
* In the opinion of the investigator has a risk of non-compliance with study procedures, or cannot read, understand, or complete study related materials, particularly the informed consent.
* Known allergy to any of the tablet or capsule excipients, or history of drug or other allergy, which, in the opinion of the responsible study physician, contraindicates participation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2007-08-17 (Actual); Primary Completion 2008-06-05 (Actual); Study Completion 2008-06-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (136):
- United States (57):
  - GSK Investigational Site, Mesa, Arizona
  - GSK Investigational Site, Artesia, California
  - GSK Investigational Site, Buena Park, California
  - GSK Investigational Site, Fresno, California
  - GSK Investigational Site, Greenbrae, California
  - GSK Investigational Site, La Jolla, California
  - GSK Investigational Site, Norwalk, California
  - GSK Investigational Site, Petaluma, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, San Mateo, California
  - GSK Investigational Site, Santa Ana, California
  - GSK Investigational Site, Tarzana, California
  - GSK Investigational Site, Torrance, California
  - GSK Investigational Site, Deland/Florida, Florida
  - GSK Investigational Site, Hollywood, Florida
  - GSK Investigational Site, Jacksonville/Florida, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Ocoee/Florida, Florida
  - GSK Investigational Site, Saint Cloud, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Bloomingdale, Illinois
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Oak Brook, Illinois
  - GSK Investigational Site, South Bend, Indiana
  - GSK Investigational Site, Lafayette, Louisiana
  - GSK Investigational Site, Lake Charles, Louisiana
  - GSK Investigational Site, Oxon Hill, Maryland
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Gulfport, Mississippi
  - GSK Investigational Site, Jackson, Mississippi
  - GSK Investigational Site, Kosciusko, Mississippi
  - GSK Investigational Site, Rolling Fork, Mississippi
  - GSK Investigational Site, Chesterfield, Missouri
  - GSK Investigational Site, Saint Louis/Missouri, Missouri
  - GSK Investigational Site, Henderson, Nevada
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Clifton, New Jersey
  - GSK Investigational Site, Albuquerque, New Mexico
  - GSK Investigational Site, Commack, New York
  - GSK Investigational Site, Ithaca, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Asheboro/North Carolina, North Carolina
  - GSK Investigational Site, Canal Fulton, Ohio
  - GSK Investigational Site, Bensalem/Pennsylvania, Pennsylvania
  - GSK Investigational Site, West Chester, Pennsylvania
  - GSK Investigational Site, Manning, South Carolina
  - GSK Investigational Site, Simpsonville, South Carolina
  - GSK Investigational Site, Athens/Tennessee, Tennessee
  - GSK Investigational Site, Corpus Christi, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Harlingen/Texas, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Midland, Texas
  - GSK Investigational Site, San Anonio, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Burke, Virginia
  - GSK Investigational Site, Bellevue, Washington
- Canada (11):
  - GSK Investigational Site, Langley, British Columbia
  - GSK Investigational Site, Bathurst, New Brunswick
  - GSK Investigational Site, Bay Roberts, Newfoundland and Labrador
  - GSK Investigational Site, Brampton, Ontario
  - GSK Investigational Site, Mississauga, Ontario
  - GSK Investigational Site, Oakville, Ontario
  - GSK Investigational Site, Ottawa, Ontario
  - GSK Investigational Site, Thornhill, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, L'Ancienne-Lorette, Quebec
  - GSK Investigational Site, Québec
- Czechia (2):
  - GSK Investigational Site, Brno
  - GSK Investigational Site, Prague
- Estonia (3):
  - GSK Investigational Site, Pärnu
  - GSK Investigational Site, Tallinn
  - GSK Investigational Site, Tartu
- Germany (23):
  - GSK Investigational Site, Allmendingen, Baden-Wurttemberg
  - GSK Investigational Site, Wangen, Baden-Wurttemberg
  - GSK Investigational Site, Großheirath, Bavaria
  - GSK Investigational Site, Hohenau, Bavaria
  - GSK Investigational Site, Künzing, Bavaria
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Parsberg, Bavaria
  - GSK Investigational Site, Ruhmannsfelden, Bavaria
  - GSK Investigational Site, Sulzbach-Rosenberg, Bavaria
  - GSK Investigational Site, Falkensee, Brandenburg
  - GSK Investigational Site, Brinkum/Stuhr, Lower Saxony
  - GSK Investigational Site, Einbeck, Lower Saxony
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Lüneburg, Lower Saxony
  - GSK Investigational Site, Tostedt, Lower Saxony
  - GSK Investigational Site, Haßloch, Rhineland-Palatinate
  - GSK Investigational Site, Ingelheim, Rhineland-Palatinate
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Freital, Saxony
  - GSK Investigational Site, Schmiedeberg, Saxony
  - GSK Investigational Site, Wolmirstedt, Saxony-Anhalt
  - GSK Investigational Site, Lübeck, Schleswig-Holstein
  - GSK Investigational Site, Berlin
- Greece (2):
  - GSK Investigational Site, Athens
  - GSK Investigational Site, Thessaloniki
- India (4):
  - GSK Investigational Site, Bangalore
  - GSK Investigational Site, Chennai
  - GSK Investigational Site, Mumbai
  - GSK Investigational Site, Pune
- Lithuania (2):
  - GSK Investigational Site, Kaunas
  - GSK Investigational Site, Vilnius
- Mexico (4):
  - GSK Investigational Site, Guadalajara, Jalisco
  - GSK Investigational Site, Cuernavaca, Morelos
  - GSK Investigational Site, Mérida, Yucatán
  - GSK Investigational Site, Durango
- GSK Investigational Site, Rotorua, New Zealand
- Poland (4):
  - GSK Investigational Site, Bydgoszcz
  - GSK Investigational Site, Porąbka
  - GSK Investigational Site, Siemianowice Śląskie
  - GSK Investigational Site, Wroclaw
- Puerto Rico (6):
  - GSK Investigational Site, Aibonito/Puerto Rico, Puerto Rico
  - GSK Investigational Site, Trujillo Alto/Puerto Rico, Puerto Rico
  - GSK Investigational Site, Caguas
  - GSK Investigational Site, Carolina
  - GSK Investigational Site, Ponce
  - GSK Investigational Site, Rio Piedras
- Romania (4):
  - GSK Investigational Site, Arad
  - GSK Investigational Site, Brasov
  - GSK Investigational Site, Sfântu Gheorghe
  - GSK Investigational Site, Timișoara
- Russia (5):
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Saint-Peterburgh
  - GSK Investigational Site, Tomsk
  - GSK Investigational Site, Tyumen
- South Africa (5):
  - GSK Investigational Site, Lenasia South, Gauteng
  - GSK Investigational Site, Bellville
  - GSK Investigational Site, Gauteng
  - GSK Investigational Site, Parow
  - GSK Investigational Site, Roodepoort
- Ukraine (3):
  - GSK Investigational Site, Dnipropetrovsk
  - GSK Investigational Site, Kyiv
  - GSK Investigational Site, Vinnitsa

REFERENCES:
- [Derived] Sykes AP, Kemp GL, Dobbins R, O'Connor-Semmes R, Almond SR, Wilkison WO, Walker S, Kler L. Randomized efficacy and safety trial of once-daily remogliflozin etabonate for the treatment of type 2 diabetes. Diabetes Obes Metab. 2015 Jan;17(1):98-101. doi: 10.1111/dom.12393. Epub 2014 Nov 3. PMID 25238025

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 130 centers in 14 countries (9 European, 3 International countries, Canada, and the United States) during the period from 17 August 2007 to 5 June 2008.
Pre-assignment Details: A total of 822 participants with Type 2 Diabetes Mellitus who were treatment naïve, entered the 2-week screening period. Of these, 570 were screen failures. The primary reason for screening failure was the participant not meeting eligibility criteria. Out of 252 randomized participants, 250 participants received study drug.
Groups:
- Placebo: Participants received 2 placebo tablets matching for GSK189075 twice daily (BID) before breakfast and dinner and 1 placebo capsule matching for Pioglitazone once daily (QD) before breakfast for 12 weeks
- GSK189075 100 mg QD: Participants received 2 tablets of GSK189075 50 milligrams (mg) each, 1 placebo capsule matching for Pioglitazone before breakfast and 2 placebo tablets matching for GSK189075 before dinner daily for 12 weeks.
- GSK189075 250 mg QD: Participants received 2 tablets of GSK189075 125 mg each, 1 placebo capsule matching for Pioglitazone before breakfast and 2 placebo tablets matching for GSK189075 before dinner daily for 12 weeks.
- GSK189075 500 mg QD: Participants received 2 tablets of GSK189075 250 mg each, 1 placebo capsule matching for Pioglitazone before breakfast and 2 placebo tablets matching for GSK189075 before dinner daily for 12 weeks.
- GSK189075 1000 mg QD: Participants received 2 tablets of GSK189075 500 mg each, 1 placebo capsule matching for Pioglitazone before breakfast and 2 placebo tablets matching for GSK189075 before dinner daily for 12 weeks.
- GSK189075 250 mg BID: Participants received 2 tablets of GSK189075 125 mg each, 1 placebo capsule matching for Pioglitazone before breakfast and 2 tablets of GSK189075 125 mg each before dinner daily for 12 weeks.
- Pioglitazone 30 mg QD: Participants received 2 placebo tablets matching GSK189075, 1 capsule of Pioglitazone 30 mg before breakfast and 2 placebo tablets matching GSK189075 before dinner daily for 12 weeks.
Period: Overall Study
Arm/Group | Placebo | GSK189075 100 mg QD | GSK189075 250 mg QD | GSK189075 500 mg QD | GSK189075 1000 mg QD | GSK189075 250 mg BID | Pioglitazone 30 mg QD
Started | 36 | 37 | 34 | 36 | 36 | 36 | 35
Completed | 30 | 30 | 27 | 32 | 31 | 31 | 30
Not Completed | 6 | 7 | 7 | 4 | 5 | 5 | 5
Not completed — Adverse Event | 0 | 1 | 3 | 0 | 1 | 1 | 1
Not completed — Lost to Follow-up | 1 | 1 | 3 | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 1 | 2 | 0
Not completed — Withdrawal by Subject | 5 | 3 | 1 | 3 | 3 | 2 | 3
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Liver function test abnormality | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — ST depression at randomisation in ECG | 0 | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Participants received 2 placebo tablets matching for GSK189075 BID before breakfast and dinner and 1 placebo capsule matching for Pioglitazone QD before breakfast for 12 weeks
- GSK189075 100 mg QD: Participants received 2 tablets of GSK189075 50 mg each, 1 placebo capsule matching for Pioglitazone before breakfast and 2 placebo tablets matching for GSK189075 before dinner daily for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | GSK189075 100 mg QD | GSK189075 250 mg QD | GSK189075 500 mg QD | GSK189075 1000 mg QD | GSK189075 250 mg BID | Pioglitazone 30 mg QD | Total
Number analyzed (Participants) | 36 | 37 | 34 | 36 | 36 | 36 | 35 | 250
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50.6 (10.60) | 53.5 (9.35) | 54.4 (9.57) | 52.6 (10.91) | 54.5 (10.19) | 50.0 (10.21) | 53.2 (10.35) | 52.7 (10.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 19 | 14 | 23 | 13 | 21 | 16 | 126
  Male | 16 | 18 | 20 | 13 | 23 | 15 | 19 | 124
Race/Ethnicity, Customized [Number; unit: Participants]
  African American/African Heritage | 2 | 3 | 3 | 4 | 2 | 4 | 1 | 19
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 3
  Asian - Central/South Asian Heritage | 5 | 7 | 3 | 2 | 5 | 5 | 2 | 29
  Asian - East Asian Heritage | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Asian - South East Asian Heritage | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 3
  White - Arabic/North African Heritage | 2 | 1 | 0 | 0 | 3 | 1 | 1 | 8
  White - White/Caucasian/European Heritage | 25 | 19 | 24 | 24 | 22 | 23 | 23 | 160
  Mixed Race | 1 | 6 | 3 | 6 | 4 | 1 | 6 | 27

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Hemoglobin A1c (Glycosylated Hemoglobin) (HbA1c) at Week 12
Description: The blood samples were collected at Baseline, Week 4, Week 8 and at Week 12 (or early withdrawal). Baseline was defined as the period immediately preceding treatment with study medication (Week 0). For participants with missing Baseline assessment, the last pre-therapy value prior to the Baseline visit was used as the Baseline value. Change from Baseline was the value at Week 12 minus Baseline value. The primary analysis was performed on the Intent-to-Treat (ITT) Population with Last observation carried forward (LOCF). Adjusted mean is presented as least square (LS) mean.
Time Frame: Baseline (Week 0) and at Week 12
Population: ITT Population consisted of all randomized participants who received at least one dose of study medication, had a Baseline assessment, and had at least one corresponding on-therapy efficacy assessment. Only those participants with data available at the indicated time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percentage
Groups:
- GSK189075 100 mg QD: Participants received 2 tablets of 50 mg each, 1 placebo capsule matching for Pioglitazone before breakfast and 2 placebo tablets matching for GSK189075 before dinner daily for 12 weeks.
- GSK189075 250 mg QD: Participants received 2 tablets of 125 mg each, 1 placebo capsule matching for Pioglitazone before breakfast and 2 placebo tablets matching for GSK189075 before dinner daily for 12 weeks.
- GSK189075 500 mg QD: Participants received 2 tablets of 250 mg each, 1 placebo capsule matching for Pioglitazone before breakfast and 2 placebo tablets matching for GSK189075 before dinner daily for 12 weeks.
- GSK189075 1000 mg QD: Participants received 2 tablets of 500 mg each, 1 placebo capsule matching for Pioglitazone before breakfast and 2 placebo tablets matching for GSK189075 before dinner daily for 12 weeks.
- GSK189075 250 mg BID: Participants received 2 tablets of 125 mg each, 1 placebo capsule matching for Pioglitazone before breakfast and 2 tablets of GSK189075 125 mg each before dinner daily for 12 weeks.
- Pioglitazone 30 mg QD: Participants received 2 placebo tablets matching GSK189075, 1 capsule of 30 mg before breakfast and 2 placebo tablets matching GSK189075 before dinner daily for 12 weeks.
Arm/Group | Placebo | GSK189075 100 mg QD | GSK189075 250 mg QD | GSK189075 500 mg QD | GSK189075 1000 mg QD | GSK189075 250 mg BID | Pioglitazone 30 mg QD
Number analyzed (Participants) | 33 | 36 | 32 | 34 | 35 | 35 | 34
Percentage | -0.19 (0.141) | -0.53 (0.135) | -0.75 (0.143) | -0.53 (0.139) | -0.85 (0.137) | -0.78 (0.137) | -0.38 (0.139)
Statistical Analysis 1: Comparison: Placebo vs GSK189075 100 mg QD vs GSK189075 250 mg QD vs GSK189075 500 mg QD vs GSK189075 1000 mg QD; Test type: Other — Tukey's trend test for dose response; p = 0.003, ANCOVA — Tukey's trend test adjusts for multiplicity with statistical significance based on p-value <0.05; Change=Baseline+Treatment
Statistical Analysis 2: Comparison: Placebo vs GSK189075 100 mg QD vs GSK189075 250 mg QD vs GSK189075 500 mg QD; Test type: Other — Tukey's trend test for dose response; p = 0.047, ANCOVA — Tukey's trend test adjusts for multiplicity with statistical significance based on p-value <0.05; Change=Baseline+Treatment
Statistical Analysis 3: Comparison: Placebo vs GSK189075 100 mg QD vs GSK189075 250 mg QD; Test type: Other — Tukey's trend test for dose response; p = 0.006, ANCOVA — Tukey's trend test adjusts for multiplicity with statistical significance based on p-value <0.05; Change=Baseline+Treatment
Statistical Analysis 4: Comparison: Placebo vs GSK189075 100 mg QD; Test type: Other — Tukey's trend test for dose response; p = 0.085, ANCOVA — Tukey's trend test adjusts for multiplicity with statistical significance based on p-value <0.05; Change=Baseline+Treatment
Statistical Analysis 5: Comparison: Placebo vs GSK189075 100 mg QD; Test type: Superiority or Other; p = 0.085, ANCOVA — Pairwise comparison included for informational purposes and not controlled for multiplicity; Change=Baseline+Treatment; Mean Difference (Net) = -0.34, 95% CI 2-sided [-0.73 to 0.05]
Statistical Analysis 6: Comparison: Placebo vs GSK189075 250 mg QD; Test type: Superiority or Other; p = 0.006, ANCOVA — Pairwise comparison included for informational purposes and not controlled for multiplicity; Change=Baseline+Treatment; Mean Difference (Net) = -0.56, 95% CI 2-sided [-0.95 to -0.16]
Statistical Analysis 7: Comparison: Placebo vs GSK189075 500 mg QD; Test type: Superiority or Other; p = 0.084, ANCOVA — Pairwise comparison included for informational purposes and not controlled for multiplicity; Change=Baseline+Treatment; Mean Difference (Net) = -0.34, 95% CI 2-sided [-0.73 to 0.05]
Statistical Analysis 8: Comparison: Placebo vs GSK189075 1000 mg QD; Test type: Superiority or Other; p = 0.001, ANCOVA — Pairwise comparison included for informational purposes and not controlled for multiplicity; Change=Baseline+Treatment; Mean Difference (Net) = -0.66, 95% CI 2-sided [-1.05 to -0.28]
Statistical Analysis 9: Comparison: Placebo vs GSK189075 250 mg BID; Test type: Superiority or Other; p = 0.003, ANCOVA — Pairwise comparison included for informational purposes and not controlled for multiplicity; Change=Baseline+Treatment; Mean Difference (Net) = -0.59, 95% CI 2-sided [-0.97 to -0.20]
Statistical Analysis 10: Comparison: Placebo vs Pioglitazone 30 mg QD; Test type: Superiority or Other; p = 0.337, ANCOVA — Pairwise comparison included for informational purposes and not controlled for multiplicity; Change=Baseline+Treatment; Mean Difference (Net) = -0.19, 95% CI 2-sided [-0.58 to 0.20]

2. Secondary Outcome: Mean Change From Baseline in HbA1c at Weeks 4 and 8
Description: The blood samples were collected at Baseline, Week 4, Week 8 and at Week 12 (or early withdrawal). Baseline was defined as the period immediately preceding treatment with study medication (Week 0). For participants with missing Baseline assessment, the last pre-therapy value prior to the Baseline visit was used as the Baseline value. Change from Baseline was the value at Week 4 and 8 minus Baseline value. The primary analysis was performed on the ITT Population with LOCF.
Time Frame: Baseline (Week 0) and at Week 4 nad 8
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Placebo | GSK189075 100 mg QD | GSK189075 250 mg QD | GSK189075 500 mg QD | GSK189075 1000 mg QD | GSK189075 250 mg BID | Pioglitazone 30 mg QD
Number analyzed (Participants) | 33 | 37 | 33 | 34 | 35 | 35 | 34
Percentage
  Week 4: number analyzed (Participants) | 30 | 32 | 31 | 30 | 33 | 32 | 30
  Week 4 | -0.18 (0.523) | -0.37 (0.437) | -0.57 (0.639) | -0.40 (0.528) | -0.45 (0.601) | -0.31 (0.541) | -0.07 (0.579)
  Week 8: number analyzed (Participants) | 33 | 36 | 32 | 34 | 35 | 35 | 34
  Week 8 | -0.08 (0.943) | -0.42 (0.720) | -0.76 (0.671) | -0.60 (0.827) | -0.77 (0.660) | -0.67 (0.646) | -0.25 (0.819)

3. Secondary Outcome: Mean Change From Baseline to Week 12 in Fasting Plasma Glucose (FPG)
Description: The samples were collected at Baseline, Week 2, Week 4, Week 8, Week 12 and Week 14 (follow up). Participants were asked to be on fast for at least 8 hours prior to each study visits and collection of lab samples. Baseline was defined as the period immediately preceding treatment with study medication (Week 0). For participants with missing Baseline assessment, the last pre-therapy value prior to the Baseline visit was used as the Baseline value. Change from Baseline was the value at Week 12 minus Baseline value. The primary analysis was performed on the ITT Population with LOCF. Adjusted mean is presented as LS mean.
Time Frame: Baseline (Week 0) and at Week 12
Population: ITT Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: millimoles per liter (mmol/L)
Arm/Group | Placebo | GSK189075 100 mg QD | GSK189075 250 mg QD | GSK189075 500 mg QD | GSK189075 1000 mg QD | GSK189075 250 mg BID | Pioglitazone 30 mg QD
Number analyzed (Participants) | 33 | 36 | 33 | 34 | 35 | 35 | 34
millimoles per liter (mmol/L) | -0.50 (0.298) | -1.35 (0.286) | -1.56 (0.298) | -1.13 (0.294) | -1.45 (0.289) | -1.63 (0.289) | -1.01 (0.295)
Statistical Analysis 1: Comparison: Placebo vs GSK189075 100 mg QD; Test type: Superiority or Other; p = 0.039, ANCOVA — Pairwise comparison not controlled for multiplicity; Change=Baseline+Treatment; Mean Difference (Net) = -0.85, 95% CI 2-sided [-1.67 to -0.04]
Statistical Analysis 2: Comparison: Placebo vs GSK189075 250 mg QD; Test type: Superiority or Other; p = 0.013, ANCOVA — Pairwise comparison not controlled for multiplicity; Change=Baseline+Treatment; Mean Difference (Net) = -1.06, 95% CI 2-sided [-1.89 to -0.23]
Statistical Analysis 3: Comparison: Placebo vs GSK189075 500 mg QD; Test type: Superiority or Other; p = 0.131, ANCOVA — Pairwise comparison not controlled for multiplicity; Change=Baseline+Treatment; Mean Difference (Net) = -0.64, 95% CI 2-sided [-1.46 to 0.19]
Statistical Analysis 4: Comparison: Placebo vs GSK189075 1000 mg QD; Test type: Superiority or Other; p = 0.023, ANCOVA — Pairwise comparison not controlled for multiplicity; Change=Baseline+Treatment; Mean Difference (Net) = -0.95, 95% CI 2-sided [-1.77 to -0.13]
Statistical Analysis 5: Comparison: Placebo vs GSK189075 250 mg BID; Test type: Superiority or Other; p = 0.007, ANCOVA — Pairwise comparison not controlled for multiplicity; Change=Baseline+Treatment; Mean Difference (Net) = -1.13, 95% CI 2-sided [-1.95 to -0.32]
Statistical Analysis 6: Comparison: Placebo vs Pioglitazone 30 mg QD; Test type: Superiority or Other; p = 0.223, ANCOVA — Pairwise comparison not controlled for multiplicity; Change=Baseline+Treatment; Mean Difference (Net) = -0.51, 95% CI 2-sided [-1.34 to 0.32]

4. Secondary Outcome: Mean Change From Baseline to Week 12 in Fructosamine (Corrected)
Description: The blood samples were collected at Baseline, Week 2, Week 4, Week 8, Week 12 and Week 14 (follow up). Participants were asked to be on fast for at least 8 hours prior to each study visits and collection of lab samples. Baseline was defined as the period immediately preceding treatment with study medication (Week 0). For participants with missing Baseline assessment, the last pre-therapy value prior to the Baseline visit was used as the Baseline value. Change from Baseline was the value at Week 12 minus Baseline value. The primary analysis was performed on the ITT Population with LOCF. Adjusted mean is presented as LS mean.
Time Frame: Baseline (Week 0) and at Week 12
Population: ITT Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: micromoles per liter (µmol/L)
Arm/Group | Placebo | GSK189075 100 mg QD | GSK189075 250 mg QD | GSK189075 500 mg QD | GSK189075 1000 mg QD | GSK189075 250 mg BID | Pioglitazone 30 mg QD
Number analyzed (Participants) | 33 | 36 | 30 | 33 | 33 | 35 | 33
micromoles per liter (µmol/L) | -1.4 (6.12) | -25.5 (5.94) | -36.3 (6.44) | -31.2 (6.12) | -37.9 (6.12) | -30.9 (5.94) | -15.2 (6.18)
Statistical Analysis 1: Comparison: Placebo vs GSK189075 100 mg QD; Test type: Superiority or Other; p = 0.005, ANCOVA — Pairwise comparison not controlled for multiplicity; Change=Baseline+Treatment; Mean Difference (Net) = -24.1, 95% CI 2-sided [-40.9 to -7.4]
Statistical Analysis 2: Comparison: Placebo vs GSK189075 250 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — Pairwise comparison not controlled for multiplicity; Change=Baseline+Treatment; Mean Difference (Net) = -35.0, 95% CI 2-sided [-52.5 to -17.4]
Statistical Analysis 3: Comparison: Placebo vs GSK189075 500 mg QD; Test type: Superiority or Other; p = 0.001, ANCOVA — Pairwise comparison not controlled for multiplicity; Change=Baseline+Treatment; Mean Difference (Net) = -29.8, 95% CI 2-sided [-46.9 to -12.7]
Statistical Analysis 4: Comparison: Placebo vs GSK189075 1000 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — Pairwise comparison not controlled for multiplicity; Change=Baseline+Treatment; Mean Difference (Net) = -36.5, 95% CI 2-sided [-53.6 to -19.5]
Statistical Analysis 5: Comparison: Placebo vs GSK189075 250 mg BID; Test type: Superiority or Other; p = 0.001, ANCOVA — Pairwise comparison not controlled for multiplicity; Change=Baseline+Treatment; Mean Difference (Net) = -29.5, 95% CI 2-sided [-46.3 to -12.7]
Statistical Analysis 6: Comparison: Placebo vs Pioglitazone 30 mg QD; Test type: Superiority or Other; p = 0.114, ANCOVA — Pairwise comparison not controlled for multiplicity; Change=Baseline+Treatment; Mean Difference (Net) = -13.8, 95% CI 2-sided [-31.0 to 3.4]

5. Secondary Outcome: Number of Participants Who Were HbA1c Responders at Week 12
Description: Differences between treatment groups in the proportion of participants who achieved HbA1c targets of <=6.5% and <7% at Week 12 in the ITT population with LOCF were assessed based on a logistic regression model with terms included for treatment and Baseline HbA1c. Differences between treatment groups in the proportion of participants who achieved a clinically meaningful decreases from Baseline in HbA1c (>=0.7%) at Week 12 were assessed in the same manner.
Time Frame: Week 12
Population: ITT Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK189075 100 mg QD | GSK189075 250 mg QD | GSK189075 500 mg QD | GSK189075 1000 mg QD | GSK189075 250 mg BID | Pioglitazone 30 mg QD
Number analyzed (Participants) | 33 | 36 | 32 | 34 | 35 | 35 | 34
Participants
  Responders (<=6.5%) | 3 | 5 | 4 | 4 | 7 | 6 | 4
  Responders (<7%) | 7 | 11 | 12 | 10 | 13 | 15 | 11
  Responders (reduction>=0.7%) | 9 | 13 | 18 | 13 | 18 | 21 | 13
Statistical Analysis 1: Comparison: Placebo vs GSK189075 100 mg QD; Placebo vs GSK189075 100 mg QD: Responders (<=6.5%); Test type: Superiority or Other; p = 0.757, Regression, Logistic — Pairwise comparison not controlled for multiplicity; Odds Ratio (OR) = 1.28, 95% CI 2-sided [0.27 to 6.06]
Statistical Analysis 2: Comparison: Placebo vs GSK189075 250 mg QD; Placebo vs GSK189075 250 mg QD: Responders (<=6.5%); Test type: Superiority or Other; p = 0.580, Regression, Logistic — Pairwise comparison not controlled for multiplicity; Odds Ratio (OR) = 1.58, 95% CI 2-sided [0.31 to 8.01]
Statistical Analysis 3: Comparison: Placebo vs GSK189075 500 mg QD; Placebo vs GSK189075 500 mg QD: Responders (<=6.5%); Test type: Superiority or Other; p = 0.881, Regression, Logistic — Pairwise comparison not controlled for multiplicity; Odds Ratio (OR) = 1.13, 95% CI 2-sided [0.22 to 5.73]
Statistical Analysis 4: Comparison: Placebo vs GSK189075 1000 mg QD; Placebo vs GSK189075 1000 mg QD: Responders (<=6.5%); Test type: Superiority or Other; p = 0.382, Regression, Logistic — Pairwise comparison not controlled for multiplicity; Odds Ratio (OR) = 1.95, 95% CI 2-sided [0.44 to 8.75]
Statistical Analysis 5: Comparison: Placebo vs GSK189075 250 mg BID; Placebo vs GSK189075 250 mg BID: Responders (<=6.5%); Test type: Superiority or Other; p = 0.409, Regression, Logistic — Pairwise comparison not controlled for multiplicity; Odds Ratio (OR) = 1.90, 95% CI 2-sided [0.42 to 8.68]
Statistical Analysis 6: Comparison: Placebo vs Pioglitazone 30 mg QD; Placebo vs Pioglitazone 30 mg QD: Responders (<=6.5%); Test type: Superiority or Other; p = 0.795, Regression, Logistic — Pairwise comparison not controlled for multiplicity; Odds Ratio (OR) = 1.24, 95% CI 2-sided [0.24 to 6.29]
Statistical Analysis 7: Comparison: Placebo vs GSK189075 100 mg QD; Placebo vs GSK189075 100 mg QD: Responders (<7%); Test type: Superiority or Other; p = 0.765, Regression, Logistic — Pairwise comparison not controlled for multiplicity; Odds Ratio (OR) = 1.20, 95% CI 2-sided [0.36 to 3.95]
Statistical Analysis 8: Comparison: Placebo vs GSK189075 250 mg QD; Placebo vs GSK189075 250 mg QD: Responders (<7%); Test type: Superiority or Other; p = 0.100, Regression, Logistic — Pairwise comparison not controlled for multiplicity; Odds Ratio (OR) = 2.74, 95% CI 2-sided [0.82 to 9.09]
Statistical Analysis 9: Comparison: Placebo vs GSK189075 500 mg QD; Placebo vs GSK189075 500 mg QD: Responders (<7%); Test type: Superiority or Other; p = 0.687, Regression, Logistic — Pairwise comparison not controlled for multiplicity; Odds Ratio (OR) = 1.28, 95% CI 2-sided [0.38 to 4.30]
Statistical Analysis 10: Comparison: Placebo vs GSK189075 1000 mg QD; Placebo vs GSK189075 1000 mg QD: Responders (<7%); Test type: Superiority or Other; p = 0.409, Regression, Logistic — Pairwise comparison not controlled for multiplicity; Odds Ratio (OR) = 1.66, 95% CI 2-sided [0.50 to 5.52]
Statistical Analysis 11: Comparison: Placebo vs GSK189075 250 mg BID; Placebo vs GSK189075 250 mg BID: Responders (<7%); Test type: Superiority or Other; p = 0.086, Regression, Logistic — Pairwise comparison not controlled for multiplicity; Odds Ratio (OR) = 2.81, 95% CI 2-sided [0.86 to 9.15]
Statistical Analysis 12: Comparison: Placebo vs Pioglitazone 30 mg QD; Placebo vs Pioglitazone 30 mg QD: Responders (<7%); Test type: Superiority or Other; p = 0.369, Regression, Logistic — Pairwise comparison not controlled for multiplicity; Odds Ratio (OR) = 1.75, 95% CI 2-sided [0.52 to 5.88]
Statistical Analysis 13: Comparison: Placebo vs GSK189075 100 mg QD; Placebo vs GSK189075 100 mg QD: Responders (reduction>=0.7%); Test type: Superiority or Other; p = 0.160, Regression, Logistic — Pairwise comparison not controlled for multiplicity; Odds Ratio (OR) = 2.17, 95% CI 2-sided [0.74 to 6.40]
Statistical Analysis 14: Comparison: Placebo vs GSK189075 250 mg QD; Placebo vs GSK189075 250 mg QD: Responders (reduction>=0.7%); Test type: Superiority or Other; p = 0.014, Regression, Logistic — Pairwise comparison not controlled for multiplicity; Odds Ratio (OR) = 3.87, 95% CI 2-sided [1.31 to 11.42]
Statistical Analysis 15: Comparison: Placebo vs GSK189075 500 mg QD; Placebo vs GSK189075 250 mg QD: Responders (reduction>=0.7%); Test type: Superiority or Other; p = 0.162, Regression, Logistic — Pairwise comparison not controlled for multiplicity; Odds Ratio (OR) = 2.17, 95% CI 2-sided [0.73 to 6.44]
Statistical Analysis 16: Comparison: Placebo vs GSK189075 1000 mg QD; Placebo vs GSK189075 1000 mg QD: Responders (reduction>=0.7%); Test type: Superiority or Other; p = 0.011, Regression, Logistic — Pairwise comparison not controlled for multiplicity; Odds Ratio (OR) = 4.09, 95% CI 2-sided [1.38 to 12.17]
Statistical Analysis 17: Comparison: Placebo vs GSK189075 250 mg BID; Placebo vs GSK189075 250 mg BID: Responders (reduction>=0.7%); Test type: Superiority or Other; p = 0.003, Regression, Logistic — Pairwise comparison not controlled for multiplicity; Odds Ratio (OR) = 5.31, 95% CI 2-sided [1.79 to 15.73]
Statistical Analysis 18: Comparison: Placebo vs Pioglitazone 30 mg QD; Placebo vs Pioglitazone 30 mg QD: Responders (reduction>=0.7%); Test type: Superiority or Other; p = 0.264, Regression, Logistic — Pairwise comparison not controlled for multiplicity; Odds Ratio (OR) = 1.86, 95% CI 2-sided [0.63 to 5.49]

6. Secondary Outcome: Number of Participants Who Were Fasting Plasma Glucose (FPG) Responders at Week 12
Description: Differences between treatment groups in the proportion of participants who achieved FPG targets of <7.0 millimoles per liter (mmol/L) (126 milligrams per deciliter [mg/dL]) and <7.8 mmol/L (140 mg/dL) at Week 12 in the ITT population with LOCF were assessed based on a logistic regression model with terms included for treatment and Baseline FPG. The proportion of participants who achieved the target of <5.5 mmol/L (100 mg/dL) at Week 12 within each treatment group were summarized only. Differences between treatment groups in the proportion of participants who achieved a clinically meaningful decreases from Baseline in FPG (1.7 mmol/L [>=30 mg/dL]) at Week 12 were assessed in the same manner.
Time Frame: Week 12
Population: ITT Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK189075 100 mg QD | GSK189075 250 mg QD | GSK189075 500 mg QD | GSK189075 1000 mg QD | GSK189075 250 mg BID | Pioglitazone 30 mg QD
Number analyzed (Participants) | 33 | 36 | 33 | 34 | 35 | 35 | 34
Participants
  Responders (<7 mmol/L) | 6 | 10 | 14 | 11 | 12 | 14 | 13
  Responders (<7.8 mmol/L) | 13 | 20 | 19 | 17 | 21 | 22 | 15
  Responders (reduction >=1.7 mmol/L) | 5 | 9 | 13 | 11 | 14 | 19 | 17
Statistical Analysis 1: Comparison: Placebo vs GSK189075 100 mg QD; Placebo vs GSK189075 100 mg QD: Responders (<7 mmol/L); Test type: Superiority or Other; p = 0.480, Regression, Logistic — Pairwise comparison not controlled for multiplicity; Odds Ratio (OR) = 1.55, 95% CI 2-sided [0.46 to 5.28]
Statistical Analysis 2: Comparison: Placebo vs GSK189075 250 mg QD; Placebo vs GSK189075 250 mg QD: Responders (<7 mmol/L); Test type: Superiority or Other; p = 0.011, Regression, Logistic — Pairwise comparison not controlled for multiplicity; Odds Ratio (OR) = 4.87, 95% CI 2-sided [1.44 to 16.46]
Statistical Analysis 3: Comparison: Placebo vs GSK189075 500 mg QD; Placebo vs GSK189075 500 mg QD: Responders (<7 mmol/L); Test type: Superiority or Other; p = 0.087, Regression, Logistic — Pairwise comparison not controlled for multiplicity; Odds Ratio (OR) = 2.92, 95% CI 2-sided [0.85 to 9.96]
Statistical Analysis 4: Comparison: Placebo vs GSK189075 1000 mg QD; Placebo vs GSK189075 1000 mg QD: Responders (<7 mmol/L); Test type: Superiority or Other; p = 0.082, Regression, Logistic — Pairwise comparison not controlled for multiplicity; Odds Ratio (OR) = 2.92, 95% CI 2-sided [0.87 to 9.78]
Statistical Analysis 5: Comparison: Placebo vs GSK189075 250 mg BID; Placebo vs GSK189075 250 mg BID: Responders (<7 mmol/L); Test type: Superiority or Other; p = 0.024, Regression, Logistic — Pairwise comparison not controlled for multiplicity; Odds Ratio (OR) = 4.00, 95% CI 2-sided [1.20 to 13.27]
Statistical Analysis 6: Comparison: Placebo vs Pioglitazone 30 mg QD; Placebo vs Pioglitazone 30 mg QD: Responders (<7 mmol/L); Test type: Superiority or Other; p = 0.012, Regression, Logistic — Pairwise comparison not controlled for multiplicity; Odds Ratio (OR) = 4.85, 95% CI 2-sided [1.41 to 16.66]
Statistical Analysis 7: Comparison: Placebo vs GSK189075 100 mg QD; Placebo vs GSK189075 100 mg QD: Responders (<7.8 mmol/L); Test type: Superiority or Other; p = 0.270, Regression, Logistic — Pairwise comparison not controlled for multiplicity; Odds Ratio (OR) = 1.85, 95% CI 2-sided [0.62 to 5.54]
Statistical Analysis 8: Comparison: Placebo vs GSK189075 250 mg QD; Placebo vs GSK189075 250 mg QD: Responders (<7.8 mmol/L); Test type: Superiority or Other; p = 0.043, Regression, Logistic — Pairwise comparison not controlled for multiplicity; Odds Ratio (OR) = 3.18, 95% CI 2-sided [1.04 to 9.72]
Statistical Analysis 9: Comparison: Placebo vs GSK189075 500 mg QD; Placebo vs GSK189075 500 mg QD: Responders (<7.8 mmol/L); Test type: Superiority or Other; p = 0.169, Regression, Logistic — Pairwise comparison not controlled for multiplicity; Odds Ratio (OR) = 2.17, 95% CI 2-sided [0.72 to 6.53]
Statistical Analysis 10: Comparison: Placebo vs GSK189075 1000 mg QD; Placebo vs GSK189075 1000 mg QD: Responders (<7.8 mmol/L); Test type: Superiority or Other; p = 0.042, Regression, Logistic — Pairwise comparison not controlled for multiplicity; Odds Ratio (OR) = 3.12, 95% CI 2-sided [1.04 to 9.36]
Statistical Analysis 11: Comparison: Placebo vs GSK189075 250 mg BID; Placebo vs GSK189075 250 mg BID: Responders (<7.8 mmol/L); Test type: Superiority or Other; p = 0.020, Regression, Logistic — Pairwise comparison not controlled for multiplicity; Odds Ratio (OR) = 3.69, 95% CI 2-sided [1.23 to 11.06]
Statistical Analysis 12: Comparison: Placebo vs Pioglitazone 30 mg QD; Placebo vs Pioglitazone 30 mg QD: Responders (<7.8 mmol/L); Test type: Superiority or Other; p = 0.211, Regression, Logistic — Pairwise comparison not controlled for multiplicity; Odds Ratio (OR) = 2.04, 95% CI 2-sided [0.67 to 6.24]
Statistical Analysis 13: Comparison: Placebo vs GSK189075 100 mg QD; Placebo vs GSK189075 100 mg QD: Responders (reduction >=1.7 mmol/L); Test type: Superiority or Other; p = 0.179, Regression, Logistic — Pairwise comparison not controlled for multiplicity; Odds Ratio (OR) = 2.90, 95% CI 2-sided [0.61 to 13.75]
Statistical Analysis 14: Comparison: Placebo vs GSK189075 250 mg QD; Placebo vs GSK189075 250 mg QD: Responders (reduction >=1.7 mmol/L); Test type: Superiority or Other; p = 0.030, Regression, Logistic — Pairwise comparison not controlled for multiplicity; Odds Ratio (OR) = 4.93, 95% CI 2-sided [1.17 to 20.87]
Statistical Analysis 15: Comparison: Placebo vs GSK189075 500 mg QD; Placebo vs GSK189075 500 mg QD: Responders (reduction >=1.7 mmol/L); Test type: Superiority or Other; p = 0.142, Regression, Logistic — Pairwise comparison not controlled for multiplicity; Odds Ratio (OR) = 2.99, 95% CI 2-sided [0.69 to 12.86]
Statistical Analysis 16: Comparison: Placebo vs GSK189075 1000 mg QD; Placebo vs GSK189075 1000 mg QD: Responders (reduction >=1.7 mmol/L); Test type: Superiority or Other; p = 0.012, Regression, Logistic — Pairwise comparison not controlled for multiplicity; Odds Ratio (OR) = 6.21, 95% CI 2-sided [1.49 to 25.83]
Statistical Analysis 17: Comparison: Placebo vs GSK189075 250 mg BID; Placebo vs GSK189075 250 mg BID: Responders (reduction >=1.7 mmol/L); Test type: Superiority or Other; p < 0.001, Regression, Logistic — Pairwise comparison not controlled for multiplicity; Odds Ratio (OR) = 13.01, 95% CI 2-sided [3.14 to 54.00]
Statistical Analysis 18: Comparison: Placebo vs Pioglitazone 30 mg QD; Placebo vs Pioglitazone 30 mg QD: Responders (reduction >=1.7 mmol/L); Test type: Superiority or Other; p = 0.010, Regression, Logistic — Pairwise comparison not controlled for multiplicity; Odds Ratio (OR) = 6.60, 95% CI 2-sided [1.56 to 27.99]

7. Secondary Outcome: Mean Change From Baseline to Week 12 in Triglycerides
Description: Samples were collected at Baseline and at Week 12 (or early withdrawal). Baseline was defined as the period immediately preceding treatment with study medication (Week 0). For participants with missing Baseline assessment, the last pre-therapy value prior to the Baseline visit was used as the Baseline value. Change from Baseline was the value at Week 12 minus Baseline value. Adjusted mean is presented as LS mean.
Time Frame: Baseline (Week 0) and at Week 12
Population: ITT Population with LOCF. Only those participants with data available at the indicated time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Placebo | GSK189075 100 mg QD | GSK189075 250 mg QD | GSK189075 500 mg QD | GSK189075 1000 mg QD | GSK189075 250 mg BID | Pioglitazone 30 mg QD
Number analyzed (Participants) | 32 | 34 | 28 | 33 | 31 | 30 | 32
mmol/L | -0.01 (0.142) | 0.19 (0.138) | -0.32 (0.152) | -0.16 (0.140) | -0.05 (0.144) | -0.18 (0.147) | -0.37 (0.142)
Statistical Analysis 1: Comparison: Placebo vs GSK189075 100 mg QD; Test type: Superiority or Other; p = 0.318, ANCOVA — Pairwise comparison not controlled for multiplicity; Change = Baseline + Treatment; Mean Difference (Net) = 0.20, 95% CI 2-sided [-0.19 to 0.59]
Statistical Analysis 2: Comparison: Placebo vs GSK189075 250 mg QD; Test type: Superiority or Other; p = 0.131, ANCOVA — Pairwise comparison not controlled for multiplicity; Change = Baseline + Treatment; Mean Difference (Net) = -0.32, 95% CI 2-sided [-0.73 to 0.10]
Statistical Analysis 3: Comparison: Placebo vs GSK189075 500 mg QD; Test type: Superiority or Other; p = 0.452, ANCOVA — Pairwise comparison not controlled for multiplicity; Change = Baseline + Treatment; Mean Difference (Net) = -0.15, 95% CI 2-sided [-0.54 to 0.24]
Statistical Analysis 4: Comparison: Placebo vs GSK189075 1000 mg QD; Test type: Superiority or Other; p = 0.845, ANCOVA — Pairwise comparison not controlled for multiplicity; Change = Baseline + Treatment; Mean Difference (Net) = -0.04, 95% CI 2-sided [-0.44 to 0.36]
Statistical Analysis 5: Comparison: Placebo vs GSK189075 250 mg BID; Test type: Superiority or Other; p = 0.393, ANCOVA — Pairwise comparison not controlled for multiplicity; Change = Baseline + Treatment; Mean Difference (Net) = -0.18, 95% CI 2-sided [-0.58 to 0.23]
Statistical Analysis 6: Comparison: Placebo vs Pioglitazone 30 mg QD; Test type: Superiority or Other; p = 0.072, ANCOVA — Pairwise comparison not controlled for multiplicity; Change = Baseline + Treatment; Mean Difference (Net) = -0.36, 95% CI 2-sided [-0.76 to 0.03]

8. Secondary Outcome: Mean Change From Baseline to Week 12 in Total Cholesterol
Description: as for outcome 7
Time Frame: Baseline (Week 0) and at Week 12
Population: ITT Population with LOCF. Only those participants with data available at the indicated time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Placebo | GSK189075 100 mg QD | GSK189075 250 mg QD | GSK189075 500 mg QD | GSK189075 1000 mg QD | GSK189075 250 mg BID | Pioglitazone 30 mg QD
Number analyzed (Participants) | 32 | 34 | 28 | 33 | 31 | 30 | 32
mmol/L | -0.03 (0.127) | -0.08 (0.124) | -0.12 (0.136) | 0.10 (0.126) | -0.02 (0.129) | 0.22 (0.132) | 0.00 (0.128)
Statistical Analysis 1: Comparison: Placebo vs GSK189075 100 mg QD; Test type: Superiority or Other; p = 0.767, ANCOVA — Pairwise comparison not controlled for multiplicity; Change = Baseline + Treatment; Mean Difference (Net) = -0.05, 95% CI 2-sided [-0.40 to 0.30]
Statistical Analysis 2: Comparison: Placebo vs GSK189075 250 mg QD; Test type: Superiority or Other; p = 0.604, ANCOVA — Pairwise comparison not controlled for multiplicity; Change = Baseline + Treatment; Mean Difference (Net) = -0.10, 95% CI 2-sided [-0.46 to 0.27]
Statistical Analysis 3: Comparison: Placebo vs GSK189075 500 mg QD; Test type: Superiority or Other; p = 0.483, ANCOVA — Pairwise comparison not controlled for multiplicity; Change = Baseline + Treatment; Mean Difference (Net) = 0.13, 95% CI 2-sided [-0.23 to 0.48]
Statistical Analysis 4: Comparison: Placebo vs GSK189075 1000 mg QD; Test type: Superiority or Other; p = 0.956, ANCOVA — Pairwise comparison not controlled for multiplicity; Change = Baseline + Treatment; Mean Difference (Net) = 0.01, 95% CI 2-sided [-0.35 to 0.37]
Statistical Analysis 5: Comparison: Placebo vs GSK189075 250 mg BID; Test type: Superiority or Other; p = 0.185, ANCOVA — Pairwise comparison not controlled for multiplicity; Change = Baseline + Treatment; Mean Difference (Net) = 0.24, 95% CI 2-sided [-0.12 to 0.60]
Statistical Analysis 6: Comparison: Placebo vs Pioglitazone 30 mg QD; Test type: Superiority or Other; p = 0.863, ANCOVA — Pairwise comparison not controlled for multiplicity; Change = Baseline + Treatment; Mean Difference (Net) = 0.03, 95% CI 2-sided [-0.32 to 0.39]

9. Secondary Outcome: Mean Change From Baseline to Week 12 in Low Density Lipoprotein Cholesterol (LDL-c)
Description: Blood samples were collected at Baseline and at Week 12 (or early withdrawal). Baseline was defined as the period immediately preceding treatment with study medication (Week 0). For participants with missing Baseline assessment, the last pre-therapy value prior to the Baseline visit was used as the Baseline value. Change from Baseline was the value at Week 12 minus Baseline value. Adjusted mean is presented as LS mean.
Time Frame: Baseline (Week 0) and Week 12
Population: ITT Population with LOCF. Only those participants with data available at the indicated time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Placebo | GSK189075 100 mg QD | GSK189075 250 mg QD | GSK189075 500 mg QD | GSK189075 1000 mg QD | GSK189075 250 mg BID | Pioglitazone 30 mg QD
Number analyzed (Participants) | 32 | 31 | 28 | 31 | 31 | 30 | 32
mmol/L | -0.02 (0.111) | -0.17 (0.113) | -0.03 (0.119) | 0.08 (0.114) | -0.04 (0.113) | 0.23 (0.115) | 0.07 (0.112)
Statistical Analysis 1: Comparison: Placebo vs GSK189075 100 mg QD; Test type: Superiority or Other; p = 0.348, ANCOVA — Pairwise comparison not controlled for multiplicity; Change = Baseline + Treatment; Mean Difference (Net) = -0.15, 95% CI 2-sided [-0.46 to 0.16]
Statistical Analysis 2: Comparison: Placebo vs GSK189075 250 mg QD; Test type: Superiority or Other; p = 0.952, ANCOVA — Pairwise comparison not controlled for multiplicity; Change = Baseline + Treatment; Mean Difference (Net) = -0.01, 95% CI 2-sided [-0.33 to 0.31]
Statistical Analysis 3: Comparison: Placebo vs GSK189075 500 mg QD; Test type: Superiority or Other; p = 0.523, ANCOVA — Pairwise comparison not controlled for multiplicity; Change = Baseline + Treatment; Mean Difference (Net) = 0.10, 95% CI 2-sided [-0.21 to 0.42]
Statistical Analysis 4: Comparison: Placebo vs GSK189075 1000 mg QD; Test type: Superiority or Other; p = 0.889, ANCOVA — Pairwise comparison not controlled for multiplicity; Change = Baseline + Treatment; Mean Difference (Net) = -0.02, 95% CI 2-sided [-0.34 to 0.29]
Statistical Analysis 5: Comparison: Placebo vs GSK189075 250 mg BID; Test type: Superiority or Other; p = 0.124, ANCOVA — Pairwise comparison not controlled for multiplicity; Change = Baseline + Treatment; Mean Difference (Net) = 0.25, 95% CI 2-sided [-0.07 to 0.56]
Statistical Analysis 6: Comparison: Placebo vs Pioglitazone 30 mg QD; Test type: Superiority or Other; p = 0.581, ANCOVA — Pairwise comparison not controlled for multiplicity; Change = Baseline + Treatment; Mean Difference (Net) = 0.09, 95% CI 2-sided [-0.22 to 0.40]

10. Secondary Outcome: Mean Change From Baseline to Week 12 in High Density Lipoprotein Cholesterol (HDL-c)
Description: as for outcome 9
Time Frame: Baseline (Week 0) and Week 12
Population: ITT Population with LOCF. Only those participants with data available at the indicated time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Placebo | GSK189075 100 mg QD | GSK189075 250 mg QD | GSK189075 500 mg QD | GSK189075 1000 mg QD | GSK189075 250 mg BID | Pioglitazone 30 mg QD
Number analyzed (Participants) | 32 | 34 | 28 | 33 | 31 | 30 | 32
mmol/L | -0.02 (0.027) | 0.00 (0.026) | 0.02 (0.028) | 0.06 (0.026) | 0.05 (0.027) | 0.04 (0.027) | 0.09 (0.026)
Statistical Analysis 1: Comparison: Placebo vs GSK189075 100 mg QD; Test type: Superiority or Other; p = 0.518, ANCOVA — Pairwise comparison not controlled for multiplicity; Change = Baseline + Treatment; Mean Difference (Net) = 0.02, 95% CI 2-sided [-0.05 to 0.10]
Statistical Analysis 2: Comparison: Placebo vs GSK189075 250 mg QD; Test type: Superiority or Other; p = 0.352, ANCOVA — Pairwise comparison not controlled for multiplicity; Change = Baseline + Treatment; Mean Difference (Net) = 0.04, 95% CI 2-sided [-0.04 to 0.11]
Statistical Analysis 3: Comparison: Placebo vs GSK189075 500 mg QD; Test type: Superiority or Other; p = 0.026, ANCOVA — Pairwise comparison not controlled for multiplicity; Change = Baseline + Treatment; Mean Difference (Net) = 0.08, 95% CI 2-sided [0.01 to 0.16]
Statistical Analysis 4: Comparison: Placebo vs GSK189075 1000 mg QD; Test type: Superiority or Other; p = 0.069, ANCOVA — Pairwise comparison not controlled for multiplicity; Change = Baseline + Treatment; Mean Difference (Net) = 0.07, 95% CI 2-sided [-0.01 to 0.14]
Statistical Analysis 5: Comparison: Placebo vs GSK189075 250 mg BID; Test type: Superiority or Other; p = 0.154, ANCOVA — Pairwise comparison not controlled for multiplicity; Change = Baseline + Treatment; Mean Difference (Net) = 0.06, 95% CI 2-sided [-0.02 to 0.13]
Statistical Analysis 6: Comparison: Placebo vs Pioglitazone 30 mg QD; Test type: Superiority or Other; p = 0.005, ANCOVA — Pairwise comparison not controlled for multiplicity; Change = Baseline + Treatment; Mean Difference (Net) = 0.11, 95% CI 2-sided [0.03 to 0.18]

11. Secondary Outcome: Mean Change From Baseline to Week 12 in LDL-c/HDL-c Ratio
Description: as for outcome 9
Time Frame: Baseline (Week 0) and Week 12
Population: ITT Population with LOCF. Only those participants with data available at the indicated time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Ratio
Arm/Group | Placebo | GSK189075 100 mg QD | GSK189075 250 mg QD | GSK189075 500 mg QD | GSK189075 1000 mg QD | GSK189075 250 mg BID | Pioglitazone 30 mg QD
Number analyzed (Participants) | 32 | 31 | 28 | 31 | 31 | 30 | 32
Ratio | 0.06 (0.119) | -0.19 (0.121) | -0.06 (0.127) | -0.13 (0.120) | -0.07 (0.121) | 0.10 (0.122) | -0.07 (0.120)
Statistical Analysis 1: Comparison: Placebo vs GSK189075 100 mg QD; Test type: Superiority or Other; p = 0.143, ANCOVA — Pairwise comparison not controlled for multiplicity; Change = Baseline + Treatment; Mean Difference (Net) = -0.25, 95% CI 2-sided [-0.58 to 0.08]
Statistical Analysis 2: Comparison: Placebo vs GSK189075 250 mg QD; Test type: Superiority or Other; p = 0.495, ANCOVA — Pairwise comparison not controlled for multiplicity; Change = Baseline + Treatment; Mean Difference (Net) = -0.12, 95% CI 2-sided [-0.46 to 0.22]
Statistical Analysis 3: Comparison: Placebo vs GSK189075 500 mg QD; Test type: Superiority or Other; p = 0.261, ANCOVA — Pairwise comparison not controlled for multiplicity; Change = Baseline + Treatment; Mean Difference (Net) = -0.19, 95% CI 2-sided [-0.52 to 0.14]
Statistical Analysis 4: Comparison: Placebo vs GSK189075 1000 mg QD; Test type: Superiority or Other; p = 0.446, ANCOVA — Pairwise comparison not controlled for multiplicity; Change = Baseline + Treatment; Mean Difference (Net) = -0.13, 95% CI 2-sided [-0.46 to 0.20]
Statistical Analysis 5: Comparison: Placebo vs GSK189075 250 mg BID; Test type: Superiority or Other; p = 0.783, ANCOVA — Pairwise comparison not controlled for multiplicity; Change = Baseline + Treatment; Mean Difference (Net) = 0.05, 95% CI 2-sided [-0.29 to 0.38]
Statistical Analysis 6: Comparison: Placebo vs Pioglitazone 30 mg QD; Test type: Superiority or Other; p = 0.454, ANCOVA — Pairwise comparison not controlled for multiplicity; Change = Baseline + Treatment; Mean Difference (Net) = -0.13, 95% CI 2-sided [-0.46 to 0.21]

12. Secondary Outcome: Mean Change From Baseline to Week 12 in Total Cholesterol/HDL-c Ratio
Description: as for outcome 9
Time Frame: Baseline (Week 0) and Week 12
Population: ITT Population with LOCF. Only those participants with data available at the indicated time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Ratio
Arm/Group | Placebo | GSK189075 100 mg QD | GSK189075 250 mg QD | GSK189075 500 mg QD | GSK189075 1000 mg QD | GSK189075 250 mg BID | Pioglitazone 30 mg QD
Number analyzed (Participants) | 32 | 34 | 28 | 33 | 31 | 30 | 32
Ratio | 0.14 (0.146) | -0.05 (0.142) | -0.20 (0.156) | -0.22 (0.144) | -0.09 (0.149) | 0.01 (0.151) | -0.26 (0.147)
Statistical Analysis 1: Comparison: Placebo vs GSK189075 100 mg QD; Test type: Superiority or Other; p = 0.363, ANCOVA — Pairwise comparison not controlled for multiplicity; Change = Baseline + Treatment; Mean Difference (Net) = -0.19, 95% CI 2-sided [-0.59 to 0.22]
Statistical Analysis 2: Comparison: Placebo vs GSK189075 250 mg QD; Test type: Superiority or Other; p = 0.111, ANCOVA — Pairwise comparison not controlled for multiplicity; Change = Baseline + Treatment; Mean Difference (Net) = -0.34, 95% CI 2-sided [-0.76 to 0.08]
Statistical Analysis 3: Comparison: Placebo vs GSK189075 500 mg QD; Test type: Superiority or Other; p = 0.080, ANCOVA — Pairwise comparison not controlled for multiplicity; Change = Baseline + Treatment; Mean Difference (Net) = -0.36, 95% CI 2-sided [-0.77 to 0.04]
Statistical Analysis 4: Comparison: Placebo vs GSK189075 1000 mg QD; Test type: Superiority or Other; p = 0.267, ANCOVA — Pairwise comparison not controlled for multiplicity; Change = Baseline + Treatment; Mean Difference (Net) = -0.23, 95% CI 2-sided [-0.64 to 0.18]
Statistical Analysis 5: Comparison: Placebo vs GSK189075 250 mg BID; Test type: Superiority or Other; p = 0.549, ANCOVA — Pairwise comparison not controlled for multiplicity; Change = Baseline + Treatment; Mean Difference (Net) = -0.13, 95% CI 2-sided [-0.54 to 0.29]
Statistical Analysis 6: Comparison: Placebo vs Pioglitazone 30 mg QD; Test type: Superiority or Other; p = 0.056, ANCOVA — Pairwise comparison not controlled for multiplicity; Change = Baseline + Treatment; Mean Difference (Net) = -0.40, 95% CI 2-sided [-0.81 to 0.01]

13. Secondary Outcome: Mean Change From Baseline to Week 12 in Body Weight
Description: Body weight measurement was taken at Baseline, Week 2, Week 4, Week 8, Week 12 and at Week 14 (follow up). Baseline was defined as the period immediately preceding treatment with study medication (Week 0). For participants with missing Baseline assessment, the last pre-therapy value prior to the Baseline visit was used as the Baseline value. Change from Baseline was the value at Week 12 minus Baseline value. Adjusted mean is presented as LS mean.
Time Frame: Baseline (Week 0) and Week 12
Population: ITT Population with LOCF.
Measure: Least Squares Mean (Standard Error); unit: kilograms
Arm/Group | Placebo | GSK189075 100 mg QD | GSK189075 250 mg QD | GSK189075 500 mg QD | GSK189075 1000 mg QD | GSK189075 250 mg BID | Pioglitazone 30 mg QD
Number analyzed (Participants) | 33 | 37 | 33 | 34 | 35 | 35 | 34
kilograms | -1.03 (0.426) | -1.52 (0.402) | -2.54 (0.425) | -2.46 (0.419) | -2.47 (0.413) | -2.11 (0.413) | 0.00 (0.419)
Statistical Analysis 1: Comparison: Placebo vs GSK189075 100 mg QD; Test type: Superiority or Other; p = 0.396, ANCOVA — Pairwise comparison not controlled for multiplicity; Change = Baseline + Treatment; Mean Difference (Net) = -0.50, 95% CI 2-sided [-1.65 to 0.66]
Statistical Analysis 2: Comparison: Placebo vs GSK189075 250 mg QD; Test type: Superiority or Other; p = 0.013, ANCOVA — Pairwise comparison not controlled for multiplicity; Change = Baseline + Treatment; Mean Difference (Net) = -1.51, 95% CI 2-sided [-2.70 to -0.33]
Statistical Analysis 3: Comparison: Placebo vs GSK189075 500 mg QD; Test type: Superiority or Other; p = 0.017, ANCOVA — Pairwise comparison not controlled for multiplicity; Change = Baseline + Treatment; Mean Difference (Net) = -1.44, 95% CI 2-sided [-2.61 to -0.26]
Statistical Analysis 4: Comparison: Placebo vs GSK189075 1000 mg QD; Test type: Superiority or Other; p = 0.015, ANCOVA — Pairwise comparison not controlled for multiplicity; Change = Baseline + Treatment; Mean Difference (Net) = -1.45, 95% CI 2-sided [-2.61 to -0.28]
Statistical Analysis 5: Comparison: Placebo vs GSK189075 250 mg BID; Test type: Superiority or Other; p = 0.069, ANCOVA — Pairwise comparison not controlled for multiplicity; Change = Baseline + Treatment; Mean Difference (Net) = -1.09, 95% CI 2-sided [-2.26 to 0.08]
Statistical Analysis 6: Comparison: Placebo vs Pioglitazone 30 mg QD; Test type: Superiority or Other; p = 0.086, ANCOVA — Pairwise comparison not controlled for multiplicity; Change = Baseline + Treatment; Mean Difference (Net) = 1.03, 95% CI 2-sided [-0.15 to 2.20]

14. Secondary Outcome: Number of Participants With Any On-therapy Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: AE was defined as any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE was defined as any untoward event resulting in death, life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, congenital anomaly/birth defect or any other situation according to medical or scientific judgment.
Time Frame: Up to Week 12
Population: Safety Population consisted of all participants who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK189075 100 mg QD | GSK189075 250 mg QD | GSK189075 500 mg QD | GSK189075 1000 mg QD | GSK189075 250 mg BID | Pioglitazone 30 mg QD
Number analyzed (Participants) | 36 | 37 | 34 | 36 | 36 | 36 | 35
Participants
  Any AEs | 8 | 15 | 20 | 11 | 21 | 20 | 12
  Any SAEs | 0 | 1 | 0 | 0 | 0 | 1 | 0

15. Secondary Outcome: Number of Participants With On-therapy Hypoglycemia
Description: Participants were provided with a Daily Glucose Monitoring Log to record glucose meter readings and to record symptoms of hypoglycemia. A separate electronic case report form (eCRF) page was provided to capture events of hypoglycemia.
Time Frame: Up to Week 12
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK189075 100 mg QD | GSK189075 250 mg QD | GSK189075 500 mg QD | GSK189075 1000 mg QD | GSK189075 250 mg BID | Pioglitazone 30 mg QD
Number analyzed (Participants) | 36 | 37 | 34 | 36 | 36 | 36 | 35
Participants | 0 | 1 | 0 | 2 | 1 | 1 | 0

16. Secondary Outcome: Number of Participants With Vital Signs of Potential Clinical Importance (PCI) at Any Time on Therapy
Description: Systolic blood pressure (SBP), diastolic blood pressure (DBP), heart rate (HR) were measured pre-dose in duplicate, after the participant has been lying quietly for 5 minutes, and then in duplicate 3 minutes after standing up. Participants were asked to refrain from smoking for at least 30 minutes prior to vital sign measurements.
Time Frame: Up to Week 12
Population: Safety Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK189075 100 mg QD | GSK189075 250 mg QD | GSK189075 500 mg QD | GSK189075 1000 mg QD | GSK189075 250 mg BID | Pioglitazone 30 mg QD
Number analyzed (Participants) | 33 | 37 | 33 | 34 | 35 | 35 | 34
Participants
  SBP, supine, low | 1 | 2 | 0 | 3 | 2 | 2 | 3
  DBP, supine, high | 0 | 0 | 0 | 0 | 0 | 1 | 0
  HR, supine, low | 1 | 0 | 0 | 0 | 1 | 0 | 1
  Orthostatic SBP, standing, low | 1 | 0 | 3 | 4 | 0 | 1 | 0
  Orthostatic DBP, standing, low | 1 | 1 | 3 | 2 | 0 | 1 | 1
  Orthostatic HR, standing, high | 4 | 5 | 6 | 5 | 5 | 7 | 5

17. Secondary Outcome: Number of Participants With Abnormal Electrocardiogram (ECG) Findings at Any Time Post-Baseline
Description: Full 12-lead ECGs were recorded at Randomization (Week 0), Week 4, and Week 12 or early withdrawal. If the QTc was >500 milliseconds on the locally read ECG recording, an additional 2 ECG recordings at 10 minute intervals were made at that visit. If the average QTc for the 3 recordings was >500 milliseconds, the participant was withdrawn from the study.
Time Frame: Up to Week 12
Population: Safety Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK189075 100 mg QD | GSK189075 250 mg QD | GSK189075 500 mg QD | GSK189075 1000 mg QD | GSK189075 250 mg BID | Pioglitazone 30 mg QD
Number analyzed (Participants) | 33 | 36 | 33 | 34 | 35 | 35 | 34
Participants | 9 | 12 | 11 | 7 | 14 | 7 | 8

18. Secondary Outcome: Number of Participants With Abnormal Chemistry Value of PCI at Any Time on Therapy
Description: Chemistry parameters: Albumin, Alkaline phosphatase, Alanine animotransferase, Aspartate aminotransferase, Total billirubin, Calcium, Carbon dioxide/Bicarbonate, Glucose, Potassium, Sodium, Phosphorus and Total protein were assessed for abnormal PCI values. Participants were instructed to fast for at least 8 hours prior to all study visits for the collection of laboratory samples. Samples were collected at Baseline, Week 2, Week 4, Week 8, Week 12 and at Week 14 (follow up).
Time Frame: Up to Week 12
Population: Safety Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK189075 100 mg QD | GSK189075 250 mg QD | GSK189075 500 mg QD | GSK189075 1000 mg QD | GSK189075 250 mg BID | Pioglitazone 30 mg QD
Number analyzed (Participants) | 33 | 37 | 33 | 34 | 35 | 35 | 34
Participants
  Albumin, low | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Alkaline phosphatase, high | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Alanine aminotransferase, high | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Aspartate aminotransferase, high | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Total bilirubin, high | 1 | 1 | 0 | 0 | 1 | 1 | 2
  Calcium, low | 0 | 1 | 3 | 0 | 0 | 2 | 0
  carbon dioxide content/Bicarbonate, low | 0 | 2 | 0 | 1 | 1 | 1 | 0
  Glucose, high | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Potassium, high | 0 | 0 | 1 | 0 | 2 | 1 | 0
  Potassium, low | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Sodium, high | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Phosphorus, high | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Total protein, high | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Total protein, low | 0 | 1 | 0 | 0 | 0 | 0 | 0

19. Secondary Outcome: Number of Participants With Abnormal Hematology Value of PCI at Any Time on Therapy
Description: Hematology parameters: Hemoglobin, Hematocrit, Platelet count and White blood cells were assessed for abnormal PCI values. Participants were instructed to fast for at least 8 hours prior to all study visits for the collection of laboratory samples. Samples were collected at Baseline, Week 2, Week 4, Week 8, Week 12 and at Week 14 (follow up).
Time Frame: Up to Week 12
Population: Safety population. Only those participants available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK189075 100 mg QD | GSK189075 250 mg QD | GSK189075 500 mg QD | GSK189075 1000 mg QD | GSK189075 250 mg BID | Pioglitazone 30 mg QD
Number analyzed (Participants) | 36 | 37 | 34 | 36 | 36 | 36 | 35
Participants
  Hemoglobin, high: number analyzed (Participants) | 33 | 37 | 33 | 34 | 35 | 35 | 34
  Hemoglobin, high | 1 | 0 | 0 | 1 | 2 | 0 | 0
  Hemoglobin, low: number analyzed (Participants) | 33 | 37 | 33 | 34 | 35 | 35 | 34
  Hemoglobin, low | 2 | 0 | 0 | 0 | 0 | 0 | 1
  Hematocrit, high: number analyzed (Participants) | 33 | 37 | 33 | 34 | 35 | 35 | 34
  Hematocrit, high | 1 | 0 | 0 | 1 | 2 | 0 | 0
  Hematocrit, low: number analyzed (Participants) | 33 | 37 | 33 | 34 | 35 | 35 | 34
  Hematocrit, low | 1 | 2 | 0 | 0 | 0 | 0 | 0
  Platelet count, high: number analyzed (Participants) | 33 | 37 | 33 | 33 | 35 | 35 | 34
  Platelet count, high | 0 | 0 | 0 | 0 | 0 | 2 | 0
  Platelet count, low: number analyzed (Participants) | 33 | 37 | 33 | 33 | 35 | 35 | 34
  Platelet count, low | 1 | 0 | 0 | 0 | 1 | 0 | 0
  White blood cell count, low: number analyzed (Participants) | 33 | 37 | 33 | 34 | 35 | 35 | 34
  White blood cell count, low | 0 | 0 | 0 | 0 | 1 | 0 | 1

ADVERSE EVENTS:
Time Frame: AEs were reported up to Week 14
Description: Safety Population was used for reporting all AEs
Arm/Group | Placebo | GSK189075 100 mg QD | GSK189075 250 mg QD | GSK189075 500 mg QD | GSK189075 1000 mg QD | GSK189075 250 mg BID | Pioglitazone 30 mg QD
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/37 | 0/34 | 0/36 | 0/36 | 0/36 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/36 | 1/37 | 0/34 | 0/36 | 0/36 | 1/36 | 0/35
Other Adverse Events (participants affected / at risk) | 3/36 | 9/37 | 11/34 | 6/36 | 17/36 | 7/36 | 7/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=36) | GSK189075 100 mg QD (N=37) | GSK189075 250 mg QD (N=34) | GSK189075 500 mg QD (N=36) | GSK189075 1000 mg QD (N=36) | GSK189075 250 mg BID (N=36) | Pioglitazone 30 mg QD (N=35)
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Scapula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=36) | GSK189075 100 mg QD (N=37) | GSK189075 250 mg QD (N=34) | GSK189075 500 mg QD (N=36) | GSK189075 1000 mg QD (N=36) | GSK189075 250 mg BID (N=36) | Pioglitazone 30 mg QD (N=35)
Urinary tract infection (Infections and infestations) | 0 | 2 | 1 | 1 | 4 | 2 | 2
Influenza (Infections and infestations) | 0 | 2 | 2 | 2 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 3 | 0 | 0 | 0 | 1 | 3
Vaginal infection (Infections and infestations) | 0 | 1 | 0 | 1 | 2 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1 | 0 | 2 | 0 | 0
Headache (Nervous system disorders) | 0 | 4 | 2 | 2 | 3 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 4 | 0 | 2 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 3 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 2 | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.